CLINICAL TRIAL: NCT04448080
Title: Topical Anesthesia vs. Analgosedation and Pain in Micropulse Transscleral Glaucoma Treatment
Brief Title: Comparison of Topical Anesthesia and Analgosedation in Micropulse Transscleral Glaucoma Treatment
Acronym: TAPMP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP MP3
Record Dates: First submitted 2020-06-08; First posted 2020-06-25 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Micropulse Transscleral Treatment for Glaucoma; Pain
MeSH Terms: conditions — Glaucoma; Pain

STUDY DESIGN:
Intervention Model Description: This is a randomised, non-blinded, controlled clinical study comparing two types of anesthesia for MicroPulse Transscleral Laser Treatment for Glaucoma
Masking Description: non
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Anesthesia (Experimental): topical tetracaine eye drops (3 times, given in 1 minute intervals) followed by topical Xylocaine 2% Gel (alcohol-free formulation), given in 1 minute intervals for a total of 5 minutes
  Interventions: Device: Micropulse Transscleral Laser Therapy for Glaucoma (MP-TLT)
- Analgosedation (Active Comparator): Remifentanil 1mg i.v., and, Thiopental i.v., adapted to patients' weight, age, and hepatic and renal function; usually, a bolus of 150-250mg
  Interventions: Device: Micropulse Transscleral Laser Therapy for Glaucoma (MP-TLT)

INTERVENTIONS:
Device: Micropulse Transscleral Laser Therapy for Glaucoma (MP-TLT) — Intraocular pressure will be lowered by Micropulse Transscleral Laser Therapy for Glaucoma (MP-TLT) in patients with a diagnosis of glaucoma

SUMMARY:
Topical Anesthesia will be compared to Analgosedation for pain control in Micropulse Transscleral Laser Treatment for Glaucoma (MP-TLT).

DETAILED DESCRIPTION:
For a patient, the perspective of a surgical treatment can mean both, hope, and anxiety. In particular the fear of pain during and after surgery can cause tremendous anxiety. In addition, possible side effects of general anesthesia and sedation should be considered, in particular, in patients with multiple comorbidities. The investigators want to help patients to cope with their anxiety and, in addition, minimize risks of surgical procedures including side effects of anesthesia. With this project, the investigators aim to investigate whether topical anesthesia - often used in ophthalmologic surgical procedures - can sufficiently control pain during and after a glaucoma laser procedure compared to intravenous analgosedation. As primary objective, the effectiveness in pain control of analgosedation and topical anesthesia in MP-TLT will be compared. As secondary objective, the effect of the anesthetic protocol used on postoperative visual related quality of life will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary open angle glaucoma (POAG)
* age ≥18 years of age
* Visual acuity ≥0.6 Decimal-Snellen
* IOP ≥21 mmHg
* </=3 anti-glaucoma drug (AGD) classes

Exclusion Criteria:

* Diagnosis of cystoid macula edema (CME) observed by optical coherence tomography (OCT)
* Status post CME
* Diagnosis of epiretinal fibroplasia
* Status post other operations than uncomplicated cataract interventions
* Status post cataract operation less than 3 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pain at 1 hour postop | 1 hour postop
  Pain will be assessed by a Numerical Pain Rating Scale (0 to 10, where 0 stands for no pain, 1 to 3 mild pain, 4 to 6 moderate pain and, 7-10 severe pain.)
Pain at 6 hours postop | 6 hours postop
  Pain will be assessed by a Numerical Pain Rating Scale (0 to 10, where 0 stands for no pain, 1 to 3 mild pain, 4 to 6 moderate pain and, 7-10 severe pain.)
Pain at 1 day postop | 1 day postop
  Pain will be assessed by a Numerical Pain Rating Scale (0 to 10, where 0 stands for no pain, 1 to 3 mild pain, 4 to 6 moderate pain and, 7-10 severe pain.)

SECONDARY OUTCOMES:
Pain at 1 week postop | 1 week postop
  Pain will be assessed by a Numerical Pain Rating Scale (0 to 10, where 0 stands for no pain, 1 to 3 mild pain, 4 to 6 moderate pain and, 7-10 severe pain.)
Pain at 1 month postop | 1 month postop
  Pain will be assessed by a Numerical Pain Rating Scale (0 to 10, where 0 stands for no pain, 1 to 3 mild pain, 4 to 6 moderate pain and, 7-10 severe pain.)
Change in Goldman-applanation intraocular pressure | at 1 month
  The change in intraocular pressure (IOP, [mmHg]) at one month compared to baseline will be computed.
Change in number of hypotensive medication | at 1 month
  The change in the number of hypotensive medication(i.e. medication which lower the intraocular pressure) at one month compared to baseline will be computed.
Change in best corrected decimal Snellen visual acuity | at 1 month
  The change in best corrected decimal Snellen visual acuity at one month compared to baseline will be computed.
visual related quality of life | at 1 month
  change in visual related quality of life at 1 month compared to baseline will be assessed by means of National Eye Institute Visual Function Questionnaire. The National Eye Institute Visual Function Questionnaire nas a minimum value of 0 and a maximum value of 100, wheras 100 means no limitions to a normal visual related quality of life (i.e. higher values represent a better outcome).

OTHER OUTCOMES:
pupil diameter | at 1 month
  change in pupil diameter at 1 month compared to baseline will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Marc Töteberg-Harms, MD, FEBO, Principal Investigator — University Hospital Zurich, Dpt. of Ophthalmology
Locations (1):
- Department of Ophthalmology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No